CLINICAL TRIAL: NCT02722395
Title: Magnetic Resonance Imaging (MRI) Solely For Liver Stereotactic Body Radiation Therapy (SBRT)
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00071159
Record Dates: First submitted 2016-03-14; First posted 2016-03-30 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Primary Liver Cancer; Metastatic Liver Cancer From Any Cancer Site
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single arm cohort study

SUMMARY:
This study is a research and development initiative established to explore the use of magnetic resonance imaging (MRI) as a tool for managing organ motion of the liver in cancer patients planning procedures for stereotactic body radiation therapy (SBRT).

DETAILED DESCRIPTION:
There is a potential role to systematically implement MRI to establish appropriate workflow of the implementation for tumor motion management in liver SBRT. Compared to CT, MRI has many significant advantages for radiotherapy planning, including superior tumor and soft-tissue contrast, flexible imaging orientation, freedom from radiation exposure and real-time imaging. MRI solely based liver SBRT will allow for more precise delineation of target volume, less uncertainties in treatment planning, better motion management, and potentially better treatment outcome

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21
* Patients with primary stage I, II, III liver cancer or metastatic tumor in the liver from any cancer site
* Signed, specific informed consent prior to study entry
* Women of child bearing potential must have a negative serum pregnancy test

Exclusion Criteria:

* Any condition for which a MRI procedure is contraindicated including presence of metallic material in the body, such as pacemakers, non- MRI compatible surgical clips, shrapnel.
* Pregnant or breast-feeding women are excluded.
* Subjects who have difficulty lying flat on their back for extended periods of time

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage I, II, III primary liver cancer Patients with metastatic liver cancer from any cancer site
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-08; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Measure average motion trajectories | During MRI approx 1 hour
Image quality, as measured by image rating | During MRI approx 1 hour
  Image quality will be measured on a scale of 1 to 5, 1 being the best.
Image quality, as measured by tumor volume | During MRI approx 1 hour
Image quality, as measured by tumor-to-live contrast to noise ratio | During MRI approx 1 hour
Planning target volume (PTV) | During MRI approx 1 hour
  PTV is defined as PTV=internal target volume (ITV) + safety margin (M)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Czito, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No